CLINICAL TRIAL: NCT00977379
Title: XERAD: Open-Label, Phase II, Randomized, Comparative, Multicentre Trial of Concurrent Whole Brain Radiation Therapy (WBRT) and Capecitabine (Xeloda®) Followed by Maintenance Capecitabine Compared With Standard WBRT in Breast Cancer Patients With Newly Diagnosed Brain Metastasis
Brief Title: A Study of Whole Brain Radiation Therapy and Capecitabine in Breast Cancer Participants With Newly Diagnosed Brain Metastasis
Acronym: XERAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to an insufficient number of participants enrolled.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21873; 2008-007349-30
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Standard of Care

ARMS (2):
- WBRT Followed by Standard of Care (Active Comparator): Participants will receive 3000 centi-Gray (cGy) WBRT in 10 single daily fractions over 12 to 14 days (300 cGy / fraction) followed by standard of care therapy at the discretion of the treating oncologist starting no earlier than 2 weeks after completion of WBRT. The participants will be followed during the treatment until the halting of standard of care for any reason (central nervous system [CNS] or extra-cranial tumor progression, unacceptable toxicity, change of therapeutic strategy, withdrawal of participant consent, or death).
  Interventions: Radiation: WBRT; Drug: Standard of Care
- WBRT+Capecitabine Followed by Capecitabine Maintenance (Experimental): Participants will receive 3000 cGy WBRT in 10 single daily fractions over 12 to 14 days (300 cGy / fraction) concurrent with capecitabine 825 milligrams per square meter (mg/m^2) orally twice daily, Days 1-14 of a 21 day cycle for 1 cycle followed by capecitabine 1000 mg/m^2 orally twice daily Days 1-14 every 21 days starting with Cycle 2, one week after completion of WBRT and continuing until the halting of capecitabine for any reason (CNS or extra-cranial progression, unacceptable toxicity, withdrawal of participant consent or death).
  Interventions: Radiation: WBRT; Drug: Capecitabine

INTERVENTIONS:
Radiation: WBRT — 3000 cGy WBRT in 10 single daily fractions over 12 to 14 days (300 cGy / fraction).
Drug: Capecitabine — 825 mg/m^2 orally twice daily, Days 1-14 of a 21 day cycle for 1 cycle followed by 1000 mg/m^2 orally twice daily Days 1-14 every 21 days starting with Cycle 2.
  Other Names: Xeloda
  Arms: WBRT+Capecitabine Followed by Capecitabine Maintenance
Drug: Standard of Care — The choice of standard of care will be at the discretion of the treating oncologist. The protocol does not specify any particular standard of care treatment.
  Arms: WBRT Followed by Standard of Care

SUMMARY:
This open-label, randomized, parallel arm study will evaluate the effect of capecitabine administered concurrently with WBRT and as maintenance therapy in participants with breast cancer and newly diagnosed brain metastases. Participants will be randomized to receive either capecitabine with 10 days standard WBRT, or WBRT alone. Maintenance therapy will follow with capecitabine or another systemic therapy in the WBRT only group.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed breast cancer with known human epidermal receptor-2 (HER2) and hormone status
* Newly diagnosed CNS metastasis with at least one brain lesion measuring greater than or equal to (>/=) 1 centimeter (cm) or two lesions measuring >/= 0.5 to less than (<) 1 cm in longest dimension
* Participant not eligible for or refusing surgery or stereotactic radiosurgery
* Eastern cooperative oncology group (EOCG) performance status 0 to 2

Exclusion Criteria:

* Prior treatment of brain metastases
* Leptomeningeal disease
* Known contra-indication to radiotherapy or magnetic resonance imaging (MRI) or capecitabine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- France (15):
  - Arras
  - Beuvry
  - Béziers
  - Bobigny
  - Dijon
  - Le Mans
  - Lille
  - Lyon
  - Montpellier
  - Nantes
  - Narbonne
  - Nice
  - Paris
  - Rouen
  - Salouël

RESULTS

PARTICIPANT FLOW:
Groups:
- WBRT Followed by Standard of Care: Participants received 3000 centi-Gray (cGy) whole brain radiation therapy (WBRT) in 10 single daily fractions over 12 to 14 days (300 cGy / fraction) followed by standard of care therapy at the discretion of the treating oncologist starting no earlier than 2 weeks after completion of WBRT. The participants were followed during the treatment until the halting of standard of care for any reason (central nervous system [CNS] or extra-cranial tumor progression, unacceptable toxicity, change of therapeutic strategy, withdrawal of participant consent, or death).
- WBRT+Capecitabine Followed by Capecitabine Maintenance: Participants received 3000 cGy WBRT in 10 single daily fractions over 12 to 14 days (300 cGy / fraction) concurrent with capecitabine 825 milligrams per square meter (mg/m^2) orally twice daily, Days 1-14 of a 21 day cycle for 1 cycle followed by capecitabine 1000 mg/m^2 orally twice daily Days 1-14 every 21 days starting with Cycle 2, one week after completion of WBRT and continuing until the halting of capecitabine for any reason (CNS or extra-cranial progression, unacceptable toxicity, withdrawal of participant consent or death).
Period: Overall Study
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Started | 12 (Randomized) | 12 (Randomized)
Treated | 12 | 11
Completed | 0 | 0
Not Completed | 12 | 12
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 7 | 9
Not completed — Premature Study Termination | 4 | 0
Not completed — Participant Moving House | 0 | 1
Not completed — Randomization Error | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants except one participant from "WBRT+Capecitabine Followed by Capecitabine Maintenance" arm who was randomized by error.
Groups:
- WBRT Followed by Standard of Care: Participants received 3000 cGy WBRT in 10 single daily fractions over 12 to 14 days (300 cGy / fraction) followed by standard of care therapy at the discretion of the treating oncologist starting no earlier than 2 weeks after completion of WBRT. The participants were followed during the treatment until the halting of standard of care for any reason (CNS or extra-cranial tumor progression, unacceptable toxicity, change of therapeutic strategy, withdrawal of participant consent, or death).
- WBRT+Capecitabine Followed by Capecitabine Maintenance: Participants received 3000 cGy WBRT in 10 single daily fractions over 12 to 14 days (300 cGy / fraction) concurrent with capecitabine 825 mg/m^2 orally twice daily, Days 1-14 of a 21 day cycle for 1 cycle followed by capecitabine 1000 mg/m^2 orally twice daily Days 1-14 every 21 days starting with Cycle 2, one week after completion of WBRT and continuing until the halting of capecitabine for any reason (CNS or extra-cranial progression, unacceptable toxicity, withdrawal of participant consent or death).
- Total: Total of all reporting groups
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (15.6) | 57.8 (13.1) | 56.2 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Objective Central Nervous System (CNS) Response, Assessed by Centralized Independent Expert According to Magnetic Resonance Imaging (MRI) - Intent-to-Treat (ITT) Population
Description: Best objective CNS response was defined as having complete response (CR) or partial response (PR) for CNS metastasis, assessed by contrast-enhanced MRI using response evaluation criteria in solid tumors (RECIST). CR: disappearance of all CNS lesions. PR: greater than or equal to (>/=) 30 percent (%) decrease in sum of longest diameters (LD) of CNS lesions taking as reference the baseline sum LD.
Time Frame: Baseline until disease progression (PD), unacceptable toxicity, withdrawal of consent, change of therapeutic strategy (for arm "WBRT Followed by Standard of Care" only), or death, whichever occurred first (up to approximately 1 year 5.5 months overall)
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
percentage of participants | 25.0 | 36.4

2. Primary Outcome: Percentage of Participants With Best Objective CNS Response, Assessed by Centralized Independent Expert According to MRI - Per-Protocol (PP) Population
Description: Best objective CNS response was defined as having CR or PR for CNS metastasis, assessed by contrast-enhanced MRI using RECIST. CR: disappearance of all CNS lesions. PR: >/=30% decrease in sum of LD of CNS lesions taking as reference the baseline sum LD.
Time Frame: Baseline until PD, unacceptable toxicity, withdrawal of consent, change of therapeutic strategy (for arm "WBRT Followed by Standard of Care" only), or death, whichever occurred first (up to approximately 1 year 5.5 months overall)
Population: PP population included all ITT population participants excluding participants with following major protocol violations: inclusion and exclusion criteria not met; intake of prohibited treatment, protocol design and/or visit dates not respected; and missing values for main criterion without premature withdrawal.
Measure: Number; unit: percentage of participants
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 10 | 9
percentage of participants | 20.0 | 33.3

3. Secondary Outcome: Percentage of Participants With Objective CNS Response at 4 Weeks After Completion of WBRT, Assessed by Centralized Independent Expert According to MRI
Description: Objective CNS response was defined as having CR or PR for CNS metastasis, assessed by contrast-enhanced MRI using RECIST. CR: disappearance of all CNS lesions. PR: >/=30% decrease in sum of LD of CNS lesions taking as reference the baseline sum LD.
Time Frame: Baseline until PD, unacceptable toxicity, withdrawal of consent, change of therapeutic strategy (for arm "WBRT Followed by Standard of Care" only), or death, whichever occurred first up to 4 weeks after completion of WBRT (up to approximately 7 weeks)
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
percentage of participants | 25.0 | 36.4

4. Secondary Outcome: Percentage of Participants With Best Objective CNS Response, Assessed by Investigator According to MRI
Description: as for outcome 2
Time Frame: as for outcome 2
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
percentage of participants | 50.0 | 54.5

5. Secondary Outcome: Percentage of Participants With Objective CNS Response at 4 Weeks After Completion of WBRT, Assessed by Centralized Independent Expert According to MRI in 3 Dimension
Description: Objective CNS response was defined as having CR or PR for CNS metastasis, assessed by 3 dimensional MRI using RECIST. CR: disappearance of all CNS lesions. PR: >/=30% decrease in sum of LD of CNS lesions taking as reference the baseline sum LD.
Time Frame: as for outcome 3
Population: The data for this outcome was not collected as per changes in planned analysis because sufficient information on the method used was not available.
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Clinical Benefit, Assessed by Investigator According to MRI
Description: Clinical benefit was defined as having CR, PR, or stable disease (SD), assessed by contrast-enhanced MRI using RECIST. CR: disappearance of all CNS lesions. PR: >/=30 % decrease in sum of LD of CNS lesions taking as reference the baseline sum LD. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as reference smallest sum LD since treatment started. PD: a 20% or greater increase in the sum of the LD of CNS lesions taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more CNS lesions and/or unequivocal progression of existing CNS lesions.
Time Frame: as for outcome 2
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
percentage of participants | 83.3 | 72.7

7. Secondary Outcome: Percentage of Participants With Objective CNS Response at 4 Weeks After Completion of WBRT, Assessed by Investigator According to MRI
Description: Objective CNS response was defined as having CR or PR for CNS metastasis, assessed by contrast-enhanced MRI using RECIST. CR: disappearance of all CNS lesions. PR: >/=30 % decrease in sum of LD of CNS lesions taking as reference the baseline sum LD.
Time Frame: as for outcome 3
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
percentage of participants | 41.7 | 27.3

8. Secondary Outcome: Duration of CNS Response, Assessed by Investigator According to MRI
Description: Duration of CNS response was defined as the time from first documented cranial CR or PR (whichever was recorded first) until the first date CNS recurrence or progression was documented as assessed by contrast-enhanced MRI according to RECIST criteria but without exam for response confirmation. CR: disappearance of all CNS lesions. PR: >/=30 % decrease in sum of LD of CNS lesions taking as reference the baseline sum LD. PD: a 20% or greater increase in the sum of the LD of CNS lesions taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more CNS lesions and/or unequivocal progression of existing CNS lesions.
Time Frame: as for outcome 2
Population: ITT population. Here, number of participants analyzed = participants having had a CR or PR during the study.
Measure: Median (Full Range); unit: months
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 6 | 6
months | 6.2 [0 to 16] | 2.6 [0 to 11]

9. Secondary Outcome: Time to CNS Progression, Assessed by Investigator According to MRI
Description: Time to CNS progression was defined as the time from start of study treatment to first documentation of PD or death due to CNS metastasis. PD was assessed by contrast-enhanced MRI according to RECIST. PD: a 20% or greater increase in the sum of the LD of CNS lesions taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more CNS lesions and/or unequivocal progression of existing CNS lesions.
Time Frame: as for outcome 2
Population: ITT population.
Measure: Median (Full Range); unit: months
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
months | 3.8 [1 to 17] | 3.4 [1 to 15]

10. Secondary Outcome: Percentage of Participants With Best Objective Extra-cranial Disease Response, Assessed by Investigator According to Computed Tomography (CT)
Description: Best objective extra-cranial response was defined as having CR or PR for extra-cranial lesions, assessed by CT using RECIST. CR: disappearance of all extra-cranial lesions. PR: >/=30 % decrease in sum of LD of extra-cranial lesions taking as reference the baseline sum LD.
Time Frame: as for outcome 2
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
percentage of participants | 0.0 | 9.1

11. Secondary Outcome: Percentage of Participants With Objective Extra-cranial Disease Response at 4 Weeks After Completion of WBRT, Assessed by Investigator According to CT
Description: Objective extra-cranial response was defined as having CR or PR for extra-cranial lesions, assessed by CT using RECIST. CR: disappearance of all extra-cranial lesions. PR: >/=30 % decrease in sum of LD of extra-cranial lesions taking as reference the baseline sum LD.
Time Frame: as for outcome 3
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
percentage of participants | 0.0 | 9.1

12. Secondary Outcome: Time to Extra-cranial Disease Progression, Assessed by Investigator According to CT
Description: Time to extra-cranial progression was defined as the time from start of study treatment to first documentation of PD or death due to extra-cranial lesions. PD was assessed by CT according to RECIST. PD: a 20% or greater increase in the sum of the LD of extra-cranial lesions taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more extra-cranial lesions and/or unequivocal progression of existing extra-cranial lesions.
Time Frame: as for outcome 2
Population: ITT population.
Measure: Median (Full Range); unit: months
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
months | 3.5 [1 to 10] | 2.7 [1 to 15]

13. Secondary Outcome: Time to Progression, Assessed by Investigator According to MRI and CT
Description: Time to progression was defined as the time from start of study treatment to first documentation of PD or death due to tumor (CNS or extra-cranial). PD was assessed by MRI or CT according to RECIST. PD: a 20% or greater increase in the sum of the LD of CNS or extra-cranial lesions taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more CNS or extra-cranial lesions and/or unequivocal progression of existing CNS or extra-cranial lesions.
Time Frame: as for outcome 2
Population: ITT population.
Measure: Median (Full Range); unit: months
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
months | 3.3 [1 to 10] | 2.7 [1 to 15]

14. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start of study treatment to date of death due to any cause. OS was assessed using Kaplan-Meier analysis.
Time Frame: Baseline until death (up to approximately 1 year 5.5 months overall)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 12 | 11
months | 9.8 [4.3 to 17.0] | 4.6 [2.3 to 8.9]

15. Secondary Outcome: Absolute Change From Baseline in Mini Mental State (MMS) Total Score
Description: MMS was an 11-question measure that tested five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. Four items were scored on a scale of 0 to 1; 1 item was scored on a scale of 0 to 2; 3 items were scored on a scale of 0 to 3; and 3 items were scored on a scale of 0 to 5. MMS total score was obtained by adding the scores of all individual items and ranged from 0 to 30, where higher scores indicate better cognitive state.
Time Frame: Baseline, Up to end of Treatment (up to 10.6 months overall)
Population: ITT population. Here, number of participants analyzed = participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Number analyzed (Participants) | 10 | 8
units on a scale | -1.5 (4.3) | 0.9 (3.2)

ADVERSE EVENTS:
Time Frame: Throughout study (up to approximately 1 year 5.5 months overall)
Description: Safety population included all participants from "WBRT Followed by Standard of Care" arm who received at least one fraction of WBRT and all participants from "WBRT+Capecitabine Followed by Capecitabine Maintenance" arm who received at least one dose of capecitabine or one fraction of WBRT.
Arm/Group | WBRT Followed by Standard of Care | WBRT+Capecitabine Followed by Capecitabine Maintenance
Serious Adverse Events (participants affected / at risk) | 6/12 | 6/11
Other Adverse Events (participants affected / at risk) | 11/12 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT Followed by Standard of Care (N=12) | WBRT+Capecitabine Followed by Capecitabine Maintenance (N=11)
Colitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT Followed by Standard of Care (N=12) | WBRT+Capecitabine Followed by Capecitabine Maintenance (N=11)
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 5
Parotid Gland Enlargement (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 6
Asthenia (General disorders) | 6 | 5
Chest Pain (General disorders) | 2 | 1
Facial Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 3
Gait Deviation (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 1 | 0
Balance Disorder (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 6
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Intracranial Pressure Increased (Nervous system disorders) | 1 | 1
Psychomotor Skills Impaired (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2
Alopecia Areata (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 2
Eyelid Oedema (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Visual Acuity Reduced (Eye disorders) | 2 | 0
Visual Impairment (Eye disorders) | 1 | 0
Escherichia Infection (Infections and infestations) | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 0
Positive Rombergism (Investigations) | 0 | 1
Weight Decreased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was prematurely terminated due to an insufficient number of participants enrolled and therefore results are only based on a small sample of breast cancer participants with newly diagnosed brain metastasis and should be considered with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.